CLINICAL TRIAL: NCT01475071
Title: Intra-individual Comparison of Efficacy and Safety of Metvix® Natural Daylight Photodynamic Therapy Versus Conventional Metvix® Photodynamic Therapy in Subject With Mild Actinic Keratoses.
Acronym: CoMet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29102
Record Dates: First submitted 2011-10-27; First posted 2011-11-21 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2016-03

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metvix and daylight (Experimental)
  Interventions: Drug: Metvix and natural daylight PDT
- Metvix and lamp (Active Comparator)
  Interventions: Drug: Metvix and conventional PDT

INTERVENTIONS:
Drug: Metvix and natural daylight PDT — Methyl aminolevulinate, cream 160mg/g.One session at baseline and a second session administration at week 12 for lesions showing non-complete response and new lesions on target area.
  Arms: Metvix and daylight
Drug: Metvix and conventional PDT — Methyl aminolevulinate, cream, 160mg/g. One session at baseline and a second session administration at week 12 for lesions showing non-complete response and new lesions on target area.
  Arms: Metvix and lamp

SUMMARY:
The main objective of this study is to compare efficacy and safety of Metvix® natural daylight photodynamic therapy with those of Metvix® conventional photodynamic therapy with Aktilite™ lamp in subjects with mild actinic keratoses (intra-individual comparison).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female above 18 years;
2. Subject with clinical diagnosis of mild AK on the face or the scalp with or without clinical diagnosis of moderate AK on the target areas (TAs);

Exclusion Criteria:

1. Subject with clinical diagnosis of at least one severe AK on TAs
2. Subject with clinical diagnosis of other skin disease (including non-melanoma skin cancer) on the TAs;
3. Subject with pigmented AK on the TAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shumack, Principal Investigator — St George Dermatology and skin Cancer Center
Locations (6):
- Australia (6):
  - Galderma Investigational site, Phillip, Australian Capital Territory
  - Galderma Investigational Site, Kogarah, New South Wales
  - Galderma Investigational site, Sydney, New South Wales
  - Galderma Investigational site, Westmead, New South Wales
  - Galderma Investigational site, Woolloongabba, Queensland
  - Galderma Investigational site, Carlton, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects recruited from March 2012 to May 2012 in private practice and clinic.
Pre-assignment Details: No significant events
Groups:
- All Subjects Enrolled: Intra-individual Comparison: all subjects have received Metvix and daylight photodynamic therapy on one side and Metvix and conventional photodynamic therapy on the other side
Period: Overall Study
Arm/Group | All Subjects Enrolled
Started | 100
Completed | 92
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects Enrolled
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 75
Region of Enrollment [Number; unit: participants]
  Australia | 100

OUTCOME MEASURES:

1. Primary Outcome: Lesion Response
Description: Percent of lesions treated at Baseline, in complete response at Week 12
Time Frame: Week12
Population: Only Per Protocol subjects are included in this analysis
Measure: Mean (Standard Deviation); unit: percentage of lesions complete response
Groups:
- Metvix and Daylight: Metvix and daylight Photodynamic Therapy
- Metvix and Lamp: Metvix and conventional Phototodynamic Therapy
Arm/Group | Metvix and Daylight | Metvix and Lamp
Number analyzed (Participants) | 90 | 90
percentage of lesions complete response | 89.2 (15.0) | 92.8 (14.1)
Statistical Analysis 1: Comparison: Metvix and Daylight vs Metvix and Lamp; The primary purpose of this study is to demonstrate the non-inferiority of Metvix and daylight compared to Metvix and the lamp in terms of lesion complete response rate; Test type: Non-Inferiority or Equivalence — Non inferiority margin of -10%; p = 0.0345, paired Student's t statistic; Mean Difference (Final Values) = -3.5, 95% CI 1-sided [lower limit -6.8], Standard Deviation 15.6

2. Primary Outcome: Pain Score
Description: Subject self assessment of pain on a scale from 0 (no pain ) to 10 (extreme pain)
Time Frame: Baseline (during procedure), assessed after procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metvix and Daylight | Metvix and Lamp
Number analyzed (Participants) | 99 | 99
units on a scale | 0.8 (1.2) | 5.7 (2.3)
Statistical Analysis 1: Comparison: Metvix and Daylight vs Metvix and Lamp; superiority of Metvix adaylight and Metvix Lamp in term of pain; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); two-sided Wilcoxon rank signed; Mean Difference (Final Values) = -4.9, Standard Deviation 2.7

ADVERSE EVENTS:
Time Frame: From baseline to study end.
Arm/Group | Metvix and Daylight | Metvix and Lamp
Serious Adverse Events (participants affected / at risk) | 9/100 | 9/100
Other Adverse Events (participants affected / at risk) | 39/100 | 59/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix and Daylight (N=100) | Metvix and Lamp (N=100)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) — not related
deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) — not related
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — not related
gastroinstestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — not related
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — not related
coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) — not related
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — not related
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) — not related
diverticulitis (Infections and infestations) | 1 (1) | 1 (1) — not related
haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) — not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix and Daylight (N=100) | Metvix and Lamp (N=100)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 6 (8) — not related
erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
pain of skin (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10)
scab (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (9)
skin reaction (Skin and subcutaneous tissue disorders) | 24 (39) | 30 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement covered by contract.